CLINICAL TRIAL: NCT00302952
Title: A Double Blind, Placebo Controlled, Phase II, Randomized Study of Lovastatin Therapy in the Treatment of Mildly Active Rheumatoid Arthritis
Brief Title: Lovastatin for the Treatment of Mildly Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment &Study Drug Expiration (Target: 40 randomized participants /arm)
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ARA02
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovastatin (Experimental): Participants are randomized to take two 40 mg lovastatin tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion. For toxicity, the dose could either be adjusted to one 40 mg lovastatin tablet or treatment could be discontinued. In addition to the active ingredient lovastatin, each tablet contained the following ingredients: microcrystalline cellulose, lactose monohydrate, magnesium stearate, and pregelatinized starch. Butylated hydroxyanisole (BHA) was added as a preservative and D&C Yellow #10, FD&C Blue #1, and Yellow #6 were added as dyes.
  Interventions: Drug: Lovastatin
- Placebo (Placebo Comparator): Participants are randomized to take two placebo tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion. For toxicity, the dose could either be adjusted to one placebo tablet or treatment could be discontinued. The placebo tablets contained microcrystalline cellulose, NF (Avicel PH 102) and Supro AA Swedish Orange Opaque Capsule Shells, Color 4188.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin — Two 40 mg lovastatin tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion
  Other Names: Altoprev; Mevacor; Mevinolin
  Arms: Lovastatin
Drug: Placebo — Two placebo tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion
  Other Names: Inactive drug (pharmacologically)
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis and a major health problem. The purpose of this study is to determine the safety and effectiveness of lovastatin for controlling inflammation in mildly active RA.

DETAILED DESCRIPTION:
RA is characterized by persistent inflammation of peripheral joints, causing pain, stiffness, swelling, and warmth. The inflammation may cause progressive joint damage and destruction, resulting in deformity and loss of function. Both traditional and biologic disease-modifying antirheumatic drugs (DMARDs) have been prescribed for RA patients to control existing inflammatory symptoms and affect long-term prognosis. However, DMARD use is expensive, and the long-term safety of DMARDs is unknown. Lovastatin is an HMG-CoA reductase inhibitor (also known as a statin) used to lower levels of cholesterol and other fats in the blood. The purpose of this study is to examine the safety and efficacy of lovastatin in controlling inflammation in individuals with RA who have mildly active RA disease despite treatment.

Participants will be randomly assigned to one of two study arms (Experimental or Placebo). There will be four study visits over 12 weeks. At each visit, a physical exam, vital signs measurement, medication history, a pregnancy test (if applicable), and blood collection will occur. Additional safety blood testing will occur at Week 2. Tender and swollen joint counts and a Physician Global Assessment will occur at study entry and Week 12. Participants will also be asked to complete self-assessments at study entry and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA as defined by 1987 American College of Rheumatology (ACR) criteria
* Functional Class I, II, or III RA as defined by 1987 ACR criteria
* Serum C-reactive protein (CRP) measurement of greater than 5 mg/L
* Mildly active disease with at least one swollen and two tender joints, but no more than six swollen and eight tender joints
* If on corticosteroids, dose must be stable and 10 mg/day prednisone (or equivalent) or less for at least 4 weeks prior to study entry
* If on DMARD, dose must be stable for at least 4 weeks (methotrexate, leflunomide, azathioprine, etanercept, adalimumab, anakinra) or at least 3 months (hydroxychloroquine, gold, or abatacept)
* Willing to use acceptable means of contraception

Exclusion Criteria:

* Serum creatinine level greater than 1.5 mg/dL
* Currently taking a statin or have taken a statin within 12 weeks of study entry
* History of an adverse reaction to a statin
* Active or recent infection within 4 weeks of study entry
* Myositis or an unexplained elevation in creatine phosphokinase (CPK)
* Joint replacement surgery within 60 days of study entry or plan to undergo joint replacement surgery during the course of the study
* Intra-articular cortisone injections within 4 weeks of study entry
* Chronic disorders other than RA affecting the joints, including systemic lupus erythematosus (SLE), psoriatic arthritis, gout, scleroderma, or known reactive arthritis (Reiter's syndrome)
* HIV infection
* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* Treatment with infliximab within 12 weeks of study entry
* Treatment with rituximab
* Treatment with medications known to be metabolized by the cytochrome P3A4 pathway. More information about this criterion can be found in the protocol.
* Require amiodarone or verapamil
* Investigational drug or treatment during the 4 weeks or seven half-lives prior to study entry
* History of alcohol abuse
* History of liver disease, current liver disease (e.g., hepatitis, cirrhosis), or abnormal liver function (AST or ALT greater than 2 times the upper limit of normal [ULN])
* Any condition that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-11-06 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Study Chair — Feinstein Institute for Medical Research NS-LIJ Health System; Betty Diamond, MD, Study Chair — Feinstein Institute for Medical Research NS-LIJ Health System
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Justus J. Fiechtner, MD, PLLC, Lansing, Michigan
  - Feinstein Institute for Medical Research NS-LIJ Health System, Manhasset, New York
  - University of Rochester, Rochester, New York
  - Carolina Bone and Joint, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Research Institute, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Abud-Mendoza C, de la Fuente H, Cuevas-Orta E, Baranda L, Cruz-Rizo J, Gonzalez-Amaro R. Therapy with statins in patients with refractory rheumatic diseases: a preliminary study. Lupus. 2003;12(8):607-11. doi: 10.1191/0961203303lu429oa. PMID 12945719
- [Background] McCarey DW, McInnes IB, Madhok R, Hampson R, Scherbakov O, Ford I, Capell HA, Sattar N. Trial of Atorvastatin in Rheumatoid Arthritis (TARA): double-blind, randomised placebo-controlled trial. Lancet. 2004 Jun 19;363(9426):2015-21. doi: 10.1016/S0140-6736(04)16449-0. PMID 15207950
- [Result] Aranow C, Cush J, Bolster MB, Striebich CC, Dall'era M, Mackay M, Olech E, Frech T, Box J, Keating R, Wasko MC, St Clair W, Kivitz A, Huang W, Ricketts P, Welch B, Callahan S, Spychala M, Boyle K, York K, Keyes-Elstein L, Goldmuntz E, Diamond B, Davidson A. A double-blind, placebo-controlled, phase II, randomized study of lovastatin therapy in the treatment of mildly active rheumatoid arthritis. Rheumatology (Oxford). 2020 Jul 1;59(7):1505-1513. doi: 10.1093/rheumatology/kez471. PMID 31628482
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY473 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY473 — ImmPort study identifier: SDY473. Participant level data is available.
- Available data/document: Study Protocol: SDY473 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY473 — ImmPort study identifier: SDY473
- Available data/document: Study summary, -design, -adverse events, -medications, -demographics, -lab tests, -mechanistic assays, -study files: SDY473 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY473 — ImmPort study identifier: SDY473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen sites in the United States participated. The first site was activated in August 2006. The first participant was randomized in November 2007 and the last participant was randomized in February 2012.
Groups:
- Lovastatin 80 mg: Participants were randomized to take two 40 mg lovastatin tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion. In addition to the active ingredient lovastatin, each tablet contained the following ingredients: microcrystalline cellulose, lactose monohydrate, magnesium stearate, and pregelatinized starch. Butylated hydroxyanisole (BHA) was added as a preservative and D&C Yellow #10, FD&C Blue #1, and Yellow #6 were added as dyes.
- Placebo: Participants were randomized to take two placebo tablets orally once daily for a total of 12 weeks in a blinded (masked) fashion. For toxicity, the dose could either be adjusted to one placebo tablet or treatment could be discontinued. The placebo tablets contained microcrystalline cellulose, NF (Avicel PH 102) and Supro AA Swedish Orange Opaque Capsule Shells, Color 4188.
Period: Overall Study
Arm/Group | Lovastatin 80 mg | Placebo
Started | 34 | 30
Started Intent-to-Treat (ITT) | 34 | 30
Completed Intent-to-Treat (ITT) | 34 | 29 (One participant did not have a baseline C-reactive Protein and was excluded from the ITT population.)
Completed | 31 | 25
Not Completed | 3 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Elevated SGOT (AST) lab value | 0 | 1

BASELINE CHARACTERISTICS:
Population: Completed Intent-to-Treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Lovastatin 80 mg | Placebo | Total
Number analyzed (Participants) | 34 | 29 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (7.1) | 52.6 (10.4) | 54.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 29 | 63
Years with Rheumatoid Arthritis at Baseline [Mean (Standard Deviation); unit: years] — Years since rheumatoid arthritis was diagnosed by a physician. This information was gathered from the medical history during the Baseline visit.
  years | 12.5 (9.6) | 11.9 (12.6) | 12.2 (11.0)
Number of Participants at Baseline Who Were Taking Methotrexate [Number; unit: Participants] — Number of participants at Baseline who were taking methotrexate prescribed by a physician. This information was gathered from the medical history during the Baseline visit.
  Participants | 20 | 16 | 36
Number of Participants at Baseline Who Were Taking an Anti-TNF Drug [Number; unit: Participants] — Number of participants at Baseline who were taking an anti-tumor necrosis factor (Anti-TNF) drug prescribed by a physician. This information was gathered from the medical history during the Baseline visit.
  Participants | 16 | 10 | 26
Number of Participants at Baseline Who Were Taking a Biologic Drug [Number; unit: Participants] — A biologic drug for the treatment of rheumatoid arthritis is a product made from a living system, that is used to decrease disease activity and to slow the progression of joint damage and includes drugs such as such as abatacept, adalimumab, or etanercept. This information was gathered from the medical history during the Baseline visit.
  Participants | 20 | 11 | 31
C-reactive Protein (CRP) Level at Baseline [Mean (Standard Deviation); unit: mg/L] — Baseline measure description: CRP is an acute phase reactant that is used to identify the presence of nonspecific inflammation. The CRP normal reference range in this study is 0-4 mg/L. An increased CRP level indicates the presence of inflammation. Reduced CRP levels could mean a decrease in inflammation.
  mg/L | 12.2 (11.4) | 12.6 (16.4) | 12.4 (13.8)
Tender Joint Count at Baseline [Mean (Standard Deviation); unit: tender joints] — The tender joint count is the number of tender joints out of the 28 examined.
  tender joints | 4.4 (2.5) | 4.8 (2.2) | 4.6 (2.4)
Swollen Joint Count at Baseline [Mean (Standard Deviation); unit: swollen joints] — The swollen joint count is the number of swollen joints out of the 28 examined.
  swollen joints | 3.5 (1.4) | 3.8 (1.6) | 3.6 (1.5)
Patient Global Assessment of Disease Activity - Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: cm] — The Patient Global Assessment of Disease Activity is a self-reported measure of perceived disease activity obtained by responding to the question "considering all the ways that your arthritis affects you, rate how you are doing on the following scale by placing a vertical mark." A vertical mark on a 10 cm line rated 0 (very well) to 10 (very bad) determines the score. The range is 0 to 10, with 10 as the highest perceived disease activity.
  cm | 3.5 (2.3) | 4.5 (1.6) | 4.0 (2.0)
Disease Activity Score Using C-reactive Protein (DAS28-CRP) [Mean (Standard Deviation); unit: scores on a scale] — The DAS28-CRP score is on a scale of 0 to 10 and indicates current activity of rheumatoid arthritis (>5.1=high disease activity; 3.2-<=5.1=moderate disease activity; <=3.2=low disease activity; <2.6=remission). The score uses a combination of four variables: 1) the number of tender joints (of the 28 that are measured); 2) the number of swollen joints (of the 28 that are measured); 3) serum C-reactive protein (CRP) in mg/L , and 4) Patient Global Assessment of Disease Activity. Using a formula, the physician determines the score.
  scores on a scale | 3.9 (0.7) | 4.2 (0.4) | 4.0 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Log Transformed C - Reactive Protein (CRP) at Day 84
Description: Blood draw for CRP, an acute phase reactant used to identify the presence of nonspecific inflammation. Change=Day 84 value minus Baseline value. Normal serum CRP reference range in this study is 0-4 mg/L (log transformed: -4.2 to 1.4). Participants with measurements for designated time points were included in analysis. An increased CRP level indicates the presence of inflammation. Reduced CRP levels could mean a decrease in inflammation.
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Intent-to-Treat with available data
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 30 | 25
mg/L | -0.4 (0.2) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Lovastatin 80 mg vs Placebo; The p-value compares Lovastatin with the Placebo treatment group. Log transformed CRP was analyzed to meet the heterogeneity assumption for ANCOVA models; Test type: Superiority or Other; p = 0.79, ANCOVA — Adjustments were made for baseline ln(CRP), baseline DAS28-CRP score, race, methotrexate use, anti-TNF use, and disease duration

2. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST) at Day 84
Description: Blood samples were taken from participants at Baseline and Day 84. Participants with measurements for designated time points included in analysis. Change=Day 84 value minus Baseline value. A positive difference reflects an increased laboratory parameter value over time; a negative difference reflects a decreased laboratory parameter value over time. Normal laboratory values depend on a subject age, gender, and the specific laboratory methods that were used to determine the lab values. Reference: http://www.merckmanuals.com/professional/appendixes/normal_laboratory_values/blood_tests_normal_values.html
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
U/L
  Alkaline Phosphatase | -3.0 (20.4) | 0.4 (15.6)
  ALT | -1.8 (10.2) | 0.7 (10.2)
  AST | -1.2 (19.7) | 0.8 (7.3)

3. Secondary Outcome: Adjusted Mean Change From Baseline in the Disease Activity Score Using C-reactive Protein (DAS28-CRP) on Day 84
Description: The DAS28-CRP score is on a scale of 0 to 10 and indicates current activity of rheumatoid arthritis (>5.1=high disease activity; 3.2-<=5.1=moderate disease activity; <=3.2=low disease activity; <2.6=remission). The score uses a combination of four variables: 1) the number of tender joints (of the 28 that are measured); 2) the number of swollen joints (of the 28 that are measured); 3) serum C-reactive protein (CRP) lab value in mg/L , and 4) Patient Global Assessment of Disease Activity. Using a formula, the physician determines the score. Participants with measurements for designated time points included in analysis.
Time Frame: Baseline (Day 0) to Day 84 (Wk 12)
Population: Intent-to-Treat with Available Data
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 31 | 25
Scores on a scale | -0.5 (0.2) | -0.5 (0.2)
Statistical Analysis 1: Comparison: Lovastatin 80 mg vs Placebo; The p-value compares Lovastatin with the Placebo treatment group; Test type: Superiority or Other; p = 0.91, ANCOVA — Adjustments were made for baseline DAS28-CRP score; ANOVA was performed on participants with a DAS28-CRP score at Day 84

4. Secondary Outcome: Percentage of Participants Meeting ACR20 Response Criteria at Day 84 (ACR: American College of Rheumatology)
Description: Patients were ACR20 Responders if they had: at least 20% improvement in both tender joint count (28 examined) and swollen joint count (28 examined), and 20% improvement in at least three of the following 5 remaining ACR core measures: • Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm) • Patient's global assessment of disease activity (VAS 100 mm) • Physician's global assessment of disease activity (VAS 100 mm) • Patient self-assessed disability (Health Assessment Questionnaire (HAQ)) score • Acute phase reactant C-reactive protein. Participants with measurements for designated time points were included in analysis.
Time Frame: Day 84 (Wk 12)
Population: Intent-to-Treat with Available Data
Measure: Number; unit: Percentage of participants
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 31 | 25
Percentage of participants | 29.0 | 40.0
Statistical Analysis 1: Comparison: Lovastatin 80 mg vs Placebo; The p-value compares Lovastatin with the Placebo treatment group; Test type: Superiority or Other; p = 0.39, Chi-squared; Difference in Percentage = -11.0, 95% CI 2-sided [-35.9 to 14.0] — The difference in percentages is calculated as Lovastatin - Placebo

5. Secondary Outcome: Adjusted Mean Change From Baseline in Serum IgM Rheumatoid Factor by ELISA (ELISA: Enzyme-linked Immunosorbent Assay)
Description: Rheumatoid factor (RF) is an antibody often present in the blood of a person with rheumatoid arthritis. In this study, a positive value for RF was 0.5 IU/mL or greater; a negative value for RF was <0.5 IU/mL. Change= Day 84 value minus Baseline value. In general, presence of the antibody indicates aggressive rheumatoid arthritis and higher risk of joint damage. Participants with measurements for designated time points included in analysis.
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Intent-to-Treat with Available Data
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 31 | 25
IU/mL | -5.4 (4.0) | 2.8 (4.5)
Statistical Analysis 1: Comparison: Lovastatin 80 mg vs Placebo; The p-value compares Lovastatin with the Placebo treatment group; Test type: Superiority or Other; p = 0.19, ANCOVA — Adjustments were made for baseline serum IgM RF by ELISA test result. In the ANCOVA model, baseline value was a covariate; therefore, an adjustment was performed

6. Secondary Outcome: Adjusted Mean Change From Baseline in Serum Anti-cyclic Citrullinated Peptide (Anti-CCP) by ELISA (ELISA: Enzyme-linked Immunosorbent Assay)
Description: Anti-CCP antibodies are autoantibodies frequently detected in the serum of individuals with rheumatoid arthritis. In this study, a positive value for anti-CCP was 8 IU/mL or greater; a negative value for anti-CCP was <8 IU/mL. Change= subtraction of Day 0 from Day 84 anti-CCP value. In general, high levels of the antibody indicate an aggressive rheumatoid arthritis and a higher risk of joint damage. Participants with measurements for designated time points included in analysis.
Time Frame: Baseline ( Day 0), Day 84 (Wk 12)
Population: Intent-to-Treat with Available Data
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 31 | 25
IU/mL | 16.3 (12.1) | -1.0 (13.5)
Statistical Analysis 1: Comparison: Lovastatin 80 mg vs Placebo; The p-value compares Lovastatin with the Placebo treatment group; Test type: Superiority or Other; p = 0.35, ANCOVA — Adjustments were made for baseline serum anti-CCP by ELISA

7. Primary Outcome: Change From Baseline in Total Bilirubin, Creatinine, BUN, Phosphorus, Calcium, and Glucose at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
mg/dL
  Total Bilirubin | 0.0 (0.2) | 0.1 (0.2)
  Creatinine | 0.0 (0.1) | 0.0 (0.1)
  BUN | -0.4 (3.2) | -0.5 (2.3)
  Phosphorus | 0.0 (0.5) | 0.0 (0.5)
  Calcium | 0.0 (0.4) | 0.0 (0.3)
  Glucose | -4.3 (16.5) | -1.2 (18.6)

8. Primary Outcome: Change From Baseline in Albumin, Total Protein, Hemoglobin, and Mean Corpuscular Hemoglobin Concentration (MCHC) at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
g/dL
  Albumin | 0.0 (0.2) | 0.1 (0.3)
  Total Protein | 0.0 (0.4) | 0.1 (0.5)
  Hemoglobin | -0.3 (0.6) | -0.3 (0.6)
  MCHC | -0.3 (0.9) | -0.4 (1.0)

9. Primary Outcome: Change From Baseline in Potassium, Sodium, Chloride, and Total CO2 at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
mmol/L
  Potassium | 0.0 (0.3) | 0.0 (0.5)
  Sodium | -0.2 (1.8) | -0.2 (2.7)
  Chloride | -0.1 (2.3) | 0.5 (3.0)
  Total CO2 | 0.7 (2.6) | -0.5 (2.3)

10. Primary Outcome: Change From Baseline in CPK at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
U/L | -2.4 (51.2) | 8.0 (54.0)

11. Primary Outcome: Change From Baseline in Counts: White Blood Cells (WBC), Neutrophils, Bands, Lymphocytes, Monocytes, Eosinophils, Basophils, Platelets, and Reticulocytes at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: 10^3/uL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
10^3/uL
  WBC | 0.1 (1.0) | -0.4 (1.3)
  Neutrophils | 0.2 (1.0) | -0.6 (1.3)
  Bands | 0.0 (0.1) | 0.0 (0.1)
  Lymphocytes | -0.1 (0.4) | 0.1 (0.8)
  Monocytes | 0.1 (0.1) | 0.0 (0.2)
  Eosinophils | 0.0 (0.1) | 0.0 (0.2)
  Basophils | 0.0 (0.0) | 0.0 (0.0)
  Platelet Count | -8.2 (34.2) | -5.6 (56.8)
  Reticulocytes | -4.7 (15.6) | 0.0 (0.0)

12. Primary Outcome: Change From Baseline in Hematocrit (Hct) at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: % of packed red blood cells by volume
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
% of packed red blood cells by volume | -0.5 (2.2) | -0.5 (2.2)

13. Primary Outcome: Change From Baseline in Red Cell Distribution Width (RDW) at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: % of mean corpuscle volume
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
% of mean corpuscle volume | -0.4 (2.0) | 0.2 (1.1)

14. Primary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH) at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
pg | -0.4 (0.7) | 0.0 (1.3)

15. Primary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV) at Day 84
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 84 (Wk 12)
Population: Safety
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Lovastatin 80 mg | Placebo
Number analyzed (Participants) | 34 | 30
fL | -0.4 (2.3) | 0.7 (3.2)

ADVERSE EVENTS:
Time Frame: Beginning of study to end of study.
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | Lovastatin 80 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/30
Other Adverse Events (participants affected / at risk) | 23/34 | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin 80 mg (N=34) | Placebo (N=30)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin 80 mg (N=34) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment was slow and the full sample size was not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No